CLINICAL TRIAL: NCT01407172
Title: Hydrogen Sulfide and Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Christopher Kevil, Associate Professor - Pathology, Louisiana State University Health Sciences Center Shreveport
Other Study IDs: H11-110
Record Dates: First submitted 2011-07-28; First posted 2011-08-02 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; Peripheral arterial disease; Hydrogen Sulfide; Gasotransmitter
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma for additional biomarker evaluation will be stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Symptomatic PAD: Patient with symptomatic PAD as defined by the presence of typical or atypical claudication symptoms or critical limb ischemia in conjunction with ABI <0.9.
- Patients without PAD: Patients without PAD as defined by ABI>0.9 and <1.3.
- Asymptomatic PAD: Patients with asymptomatic PAD as defined by ABI<0.9 but no symptoms.

SUMMARY:
This will be an observational study comparing the plasma levels of free hydrogen sulfide in patients with and without peripheral arterial disease using a novel recently published method of measuring hydrogen sulfide. The investigators will also see if there is any difference in these levels between symptomatic and asymptomatic patients. Will examine the relationship of these levels to known clinical risk factors as well as plasma nitrite and nitric oxide levels. In doing the above the investigators hope to explore the utility of free hydrogen sulfide as a biomarker for peripheral arterial disease.

Atherosclerotic peripheral arterial disease (PAD) of the lower extremities represents a significant and growing cause of morbidity and mortality. The PARTNERS study of screening ABIs in a primary care population of nearly 7000 individuals demonstrated a remarkable 29% incidence of ABI <0.9, which is the commonly accepted level of abnormal ABI diagnostic of PAD. Also of note in these patients with a new diagnosis of PAD the incidence of asymptomatic PAD was a striking 48%. The availability of a biomarker will greatly enhance the care of these patient and hopefully reduce morbidity and mortality.

The investigators believe that hydrogen sulfide (H2S), an endogenously produced gasotransmitter, holds promise as a clinically useful biomarker for PAD and may also provide a possible explanation for the paradox of asymptomatic PAD in patients with ABIs less than 0.9. To date, research regarding H2S has demonstrated that it participates in a myriad of physiological functions including vasodilatation, anti-apoptotic effects, modulation of mitochondrial respiration, and changes in vascular remodeling.

DETAILED DESCRIPTION:
The investigators will conduct an observational cohort study to evaluate H2S levels in three groups of patients:

1. Patients without PAD as defined by ABI>0.9 and <1.3.
2. Patients with asymptomatic PAD as defined by ABI<0.9 but no symptoms
3. Patient with symptomatic PAD as defined by the presence of typical or atypical claudication symptoms or critical limb ischemia in conjunction with ABI <0.9.

This will be a single center study performed at LSUHSC-Shreveport. Patients undergoing cardiac catheterization or peripheral angiogram via a major arterial approach at the LSUHSC cardiac catheterization laboratory meeting the inclusion and exclusion criteria will be eligible and given an opportunity to participate. Those providing informed consent will be interviewed for the presence of claudication symptoms, by use of the San Diego Claudication Questionnaire and the presence of known risk factors for PAD. The medical record will be reviewed for collection of baseline clinical data including known risk factors for vascular disease as well as medications etc. Ankle Brachial Index will be measured by the standard technique of non-invasive measurement of bilateral arm and ankle pressures and recorded in all patients.

Plasma free H2S level quantification via high performance liquid gas chromatography, as well as plasma nitrite levels and nitric oxide levels by chemiluminescence assay will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled at the cardiac catheterization laboratory for coronary or peripheral angiography.
2. Age > 40 years.

Exclusion Criteria:

1. Inability to provide informed consent.
2. ST elevation myocardial infarction.
3. Cardiogenic shock.
4. Non-atherosclerotic PAD (e.g. Buerger's disease).
5. Pregnant or nursing.
6. Enrolment in another clinical trial requiring use of experimental therapeutic agents.
7. ABI > 1.3(indicative of non-compressible vessel needing further evaluation to diagnose PAD), unless documented known PAD.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac catheterization or peripheral angiogram via a major arterial approach at the LSUHSC cardiac catheterization laboratory meeting the inclusion and exclusion criteria will be eligible and given an opportunity to participate.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Free plasma hydrogen sulfide levels | day 1 at enrollment only, we will not be prospectively following these levels.
  Will be evaluating plasma free hydrogen sulfide levels in the three cohorts of patients.

SECONDARY OUTCOMES:
Plasma nitrite and nitric oxide levels. | day 1 at enrollment only, we will not be prospectively following these levels.
  Will evaluate the plasma levels of nitrite and nitric oxide in the three cohorts of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kevil, PhD, Principal Investigator — LSUHSC Shreveport
Locations (1):
- LSUHSC Shreveport, Shreveport, Louisiana, United States

REFERENCES:
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Shen X, Pattillo CB, Pardue S, Bir SC, Wang R, Kevil CG. Measurement of plasma hydrogen sulfide in vivo and in vitro. Free Radic Biol Med. 2011 May 1;50(9):1021-31. doi: 10.1016/j.freeradbiomed.2011.01.025. Epub 2011 Jan 27. PMID 21276849
- [Background] Cooke JP, Wilson AM. Biomarkers of peripheral arterial disease. J Am Coll Cardiol. 2010 May 11;55(19):2017-23. doi: 10.1016/j.jacc.2009.08.090. PMID 20447524
- [Background] Calvert JW, Coetzee WA, Lefer DJ. Novel insights into hydrogen sulfide--mediated cytoprotection. Antioxid Redox Signal. 2010 May 15;12(10):1203-17. doi: 10.1089/ars.2009.2882. PMID 19769484
- [Derived] Peter EA, Shen X, Shah SH, Pardue S, Glawe JD, Zhang WW, Reddy P, Akkus NI, Varma J, Kevil CG. Plasma free H2S levels are elevated in patients with cardiovascular disease. J Am Heart Assoc. 2013 Oct 23;2(5):e000387. doi: 10.1161/JAHA.113.000387. PMID 24152982